CLINICAL TRIAL: NCT03155113
Title: Role of the Host Immunity in the Non-response to DAA Therapy
Brief Title: Role of the Host Immunity in the Non-response to Direct Anti-viral Agent (DAA) Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Carlo Ferrari, professor, Azienda Ospedaliero-Universitaria di Parma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NR-DAA-HCV
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic infection; HCV; DAA therapy; immune response
MeSH Terms: conditions — Hepatitis C, Chronic; Persistent Infection | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with chronic HCV infection (Other): Patients with chronic HCV infection to be treated with any of the available DAA (without associated PEG-IFN) in daily clinical practice.
  Intervention: Blood Drawing.Before starting therapy a blood sample will be collected from any subject.
  Interventions: Other: blood drawing

INTERVENTIONS:
Other: blood drawing — Before starting therapy a blood sample will be collected from any subject.

SUMMARY:
Anti-viral, hepatitis C virus (HCV)-specific immune T cell responses are functionally defective in patients with chronic hepatitis C and this functional impairment is believed to contribute to virus persistence. Persistent exposure to high virus loads is likely involved in the pathogenesis of T cell dysfunction. The underlying hypothesis of the project is that the level of anti-viral immune dysfunction in chronic HCV infection is a causal factor which can influence non-response to therapy.

Although the rate of response to direct anti-viral agent (DAA) therapy, in untreated, non-cirrhotic, patients is between 95% and 100%, however, the response rate is lower in specific subgroups of patients, including genotype 3 cirrhotics and patients with decompensated cirrhosis, irrespective of the infecting genotype.

Aim of the present study will be thus to understand whether non-response to therapy is associated with a wider and deeper anti-viral immune dysfunction, by comparing individual HCV-specific T cell responses in two groups of responder and non-responder patients. Characterization of protective immunity in non-responder patients could allow to identify baseline predictors of non-response to therapy to be used in the daily clinical practice.

Objective of the study will be to compare the features (intensity and quality) of the overall HCV-specific immune T cell response in patients non-responder and responder to DAA therapy. To achieve this goal, T lymphocytes (either CD4 or CD8) isolated from the peripheral blood of the patients, before starting DAA therapy, will be stimulated with HCV proteins to evaluate the capacity of those cells to expand, produce cytokines and express cytotoxic capacity.

DETAILED DESCRIPTION:
Study objective and Hypothesis The underlying hypothesis of the project is that the level of anti-viral immune dysfunction in chronic HCV infection is a causal factor which can influence non-response to therapy. However, information about the features of individual anti-viral T cell responses expressed by naïve chronic HCV patients before starting DAA therapy in relation to the subsequent outcome of treatment and their possible impact on the failure to control infection is not available. The few available results on anti-HCV immune responses in chronic HCV infection have been generated in patients treated with DAA regimens which are not included in the present guidelines without evaluation according to the outcome. Aim of the present study will be thus to understand whether non-response to therapy is associated with a wider and deeper anti-viral immune dysfunction, by comparing individual HCV-specific T cell responses in two groups of responder and non-responder patients. The assumption made is that possible defects of T cell responses associated with the failure to respond to DAA therapy should not be substantially modified by an ineffective treatment allowing to characterize the immunological background of non responder patients after the end of an ineffective cycle of therapy and to compare results with baseline pretreatment responses of naïve, viremic patients who subsequently clear the virus. A pre-treatment analysis also for non responder patients would require to enroll a huge number of naive patients in order to identify a sufficient number of non responder patients, making the study unfeasible and exceedingly long. By this strategy, recruitment will be instead very rapid because most patients enrolled at baseline are expected to be responder, while non responder patients who will be studied after the end of therapy and after an adequate wash-out period of 6 to 12 months and before starting re-treatment have already been identified in the collaborating Centers and will be readily available for the study as soon as the protocol is approved. Based on the results, possible objective of future analyses could be to characterize further at a molecular level the T cell functional defects of non-responder patients to define whether and by which strategies their correction can represent a feasible approach to induce/restore an efficient anti-viral response to complement and strengthen the effect of last generation DAA. Finally, characterization of protective immunity in non-responder patients could allow to identify baseline predictors of non-response to therapy to be used in the daily clinical practice.

Study background The rate of sustained viral response (SVR) in naïve non-cirrhotic patients treated with IFN-free DAAs is between 95% and 100%, but the response rate is lower in specific subgroups of patients, including genotype 3 cirrhotics and patients with decompensated cirrhosis, irrespective of the infecting genotype. The high efficacy of DAA-based therapies is confirmed in real-world cohorts, which show a rate of SVR only slightly lower than registration studies. Although the rate of failure to DAA therapy is quite limited (around 5%), the overall number of non-responder patients is expected to be high because of the high number of chronically HCV infected patients who need treatment. Treatment failure most frequently results in relapse and less often in on-treatment viral breakthrough. Different factors are believed to be implicated in non-response to therapy, including emergence of resistance mutations, suboptimal treatment due to incorrect genotype definition and advanced liver disease.

The role of baseline RAVs in determining treatment failure is still debated and baseline resistance testing appears to have limited clinical utility. Instead, emergence of RAVs during DAA-based regimens and its role in determining virological failure is well documented. Even if drug-resistant variants are detected in a large proportion of non-responder patients, their role in impairing treatment efficacy is however not totally clear.

The use of currently available second-generation commercial assays for HCV genotyping has reduced the risk of genotype misclassification, but the possibility of mixed infections with a percentage of different genotypes/subtypes below the sensitivity of the methods applied in the clinical practice is still a possible cause of non response to therapy due to suboptimal treatment.

Emergence of resistant strains and suboptimal treatment due to incorrect genotype detection can however explain only part of treatment failure cases and host-related factors may play a role, in particular the anti-viral immune response. Indeed, innate and adaptive immune responses are known to be deeply impaired in chronic HCV infection but very limited information is available about the possible contribution that background immune responses can give to the final outcome of DAA treatment. In contrast to PegIFN-based therapies, recent studies in DAA treated patients indicate that frequency and function of HCV-specific CD8 cells can increase under IFN-free therapies with partial reversal of their exhausted phenotype. Moreover, DAA therapy can modulate the NK cell compartment correcting the NK cell activated phenotype which is typical of chronic HCV patients. Thus, the level of baseline impairment of anti-viral immunity might influence the subsequent likelihood of immune restoration upon therapy with more chances of resistance to DAA treatment when baseline immune inhibition is deeper and wider. This hypothesis requires to be tested.

Primary Endpoints Objective of the study will be to compare intensity (total levels of anti-viral functions) and quality (multi-specificity and multi-functionality) of the overall HCV-specific T cell response in patients non-responder (with and without detectable resistance associated variants - RAVs) and responder to DAA therapy. To achieve this goal, CD4- and CD8-mediated responses will be assessed by using overlapping synthetic peptides covering the overall HCV proteome of genotype 1 in order to characterize T cell reactivity to all HCV proteins, in terms of cytokine production (IL2, IFN-g and TNF-a) and cytotoxic potential (CD107 degranulation).

* As a primary endpoint, the overall intensity of T cell responses will be assessed in responder and non responder patients; the total intensity of individual T cell reactivity will be defined by summing the different analyzed T cell parameters (cytokine production and cytotoxicity, as detected in total CD3 cells and CD4/CD8 subsets) for each individual responder and non-responder patient; the resulting values will be then compared in the two groups of patients.
* At a second level of analysis, qualitative differences in T cell reactivity between responder and non-responder patients will be assessed in terms of multi-functionality and multi-specificity of HCV-specific T cell responses, by comparing the expression of each individual function separately (IL2, IFN-g, TNF-a) and the capacity of each individual HCV protein to induce T cell responses in the two groups of patients.

Characterization of HCV-specific T cell responses.

1. To analyze global CD4+ and CD8+ reactivity against structural and non-structural HCV proteins, a comprehensive panel of overlapping 15-mer peptides covering the entire HCV (genotypes 1) sequence will be used; T cell responses will be analyzed by flow-cytometric intracellular cytokine staining (ICS) for IFN-g, IL-2 and TNF-a and for degranulation (up-regulation of CD107) in vitro (after 10 days of peptide stimulation) and by Elispot for IFN-g ex-vivo (after short-term peptide stimulation); synthetic peptide epitopes with HLA class I- and class II-restricted specificities and known to be the targets of CD8+ and CD4+ responses against different HCV-unrelated viruses and pathogens (CMV, EBV, FLU) will be used as controls.
2. To further analyze CD8+ T cell reactivity, HLA-A2/peptide dextramers containing some of the most widely recognized HLA-A2 restricted epitopes of HCV will be used in HLA-A2+ patients to quantify circulating virus-specific CD8+ cells and to measure expansion capacity by comparing dextramer-positive CD8+ cell frequencies ex-vivo and after 10 days of peptide stimulation.
3. In non-responder patients showing the emergence of resistance mutations, specific peptides corresponding to the variant sequences will be synthesized and used to analyze whether emerging mutations can influence HCV-specific T cell activation and function. For this purpose, the stimulatory effect on different T cell functions of prototype and variant peptides (cytokine production, cytotoxicity, capacity of expansion) will be compared

Secondary Endpoints

1. Analysis of additional immune populations and serum factors known to be relevant with respect to control of virus infection and modulation of T cell responses.

   * Natural Killer (NK) cell analysis: NK cell phenotype will be studied by assessing the expression of specific markers, such as CD16, NKG2A/D, TRAIL, NKP46/NKP30, Ki67, CD38/HLA-DR by flow cytometry; NK cell function will be studied by testing IFN-g/TNF-a production and CD107 degranulation upon overnight PBMC incubation with appropriate stimuli.
   * Analysis of T regulatory cell (Treg): frequency, phenotype and function will be studied on whole PBMCs co-stained with CD3, CD4, CD25, FoxP3 and CD45RA.
   * Serum concentration of cytokines, chemokines and ISG, including IL15, IL6, CXCL9, CXCL10, IFN-g and IL28, will be analyzed in patients' sera by the Luminex technology.
2. Identification of baseline predictors of non-response to DAA therapy Elucidation of the impact that the anti-viral immune response can have in non-response to therapies with or without protease inhibitors

ELIGIBILITY:
Inclusion Criteria:

* naïve HCV genotype 1 infected chronic patients (F3-F4 fibrosis stages by liver histology of fibroscan) treated with any of the available DAA (without associated PEG-IFN) in daily clinical practice:

  1. non-responder patients, enrolled and studied after identification of non-response (at least 12 weeks after end of therapy) - 50 patients
  2. responder patients, enrolled and studied before therapy - 25 patients
* male or female, age ≥ 18 years
* quantifiable plasma HCV-RNA
* F3-F4 liver fibrosis (Metavir) assessed by liver biopsy or by FibroScan™
* treatment with an optimal DAA schedule (based on EASL guidelines)
* evidence of adherence to therapy

Exclusion Criteria:

* Mixed genotype populations by deep HCV sequencing
* Non response following a non-optimal treatment schedule
* Signs or symptoms of HCC
* History of decompensated liver disease
* Co-infection with hepatitis B or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Immune T cell response | between 12 and 14 months from the beginning of the study
  Identification of specific baseline immunological features predictors of non-response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ferrari, Dr, Principal Investigator — Università degli Studi di Parma
Locations (1):
- Unit of Infectious Diseases and Hepatology, Parma, Italy

IPD SHARING:
Plan to Share IPD: No